CLINICAL TRIAL: NCT02590471
Title: Pilot Prospective Study of Two Methods of Revascularization of the Superficial Femoral Artery: Stenting in the Superficial Femoral Artery, and Stenting of the Superficial Femoral Artery, Supplemented by Fasciotomy in Hunter Channel in Patients With Steno-occlusive Lesions of Femoral-popliteal Segment TASC C, D
Brief Title: Pilot Prospective Study of Two Methods of Revascularization of the Femoral Artery (SFA): Stenting in the SFA, and Stenting of the SFA, Supplemented by Fasciotomy in Hunter Channel.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: N-RICP-467
Record Dates: First submitted 2015-10-23; First posted 2015-10-29 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Atherosclerosis of the Peripheral Artery
Keywords: Angioplasty with stenting of the superficial femoral artery; Fasciotomy in Hunter's channel; Breakage of stent
MeSH Terms: interventions — Angioplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stenting of the femoral artery. (Active Comparator): A standard endovascular exposure is carried out under local anesthesia and a lesioned arterial segment is visualized. Stenosis or artery occlusion is passed by the hydrophilic guide. During the occlusion transluminal or subintimal artery recanalization (most frequently mixed) is conduced. Then balloon angioplasty of stenosis or occlusion are carried out. After the angiographic control if necessary stent of all the extension is mounted.
  Interventions: Procedure: Angioplasty with stenting of the femoral artery
- Stenting of the femoral artery and fasciotomy. (Experimental): Under local anesthesia standard endovascular exposure is made and lesioned arterial segment is visualized. Stenosis or artery occlusion is passed by the hydrophilic guide. During the occlusion transluminal or subintimal artery recanalization (most frequently mixed) is conduced. Then balloon angioplasty of stenosis or occlusion are carried out. After the angiographic control if necessary stent of all the extension is mounted. The exposure is carried out to the distal part of superficial femoral artery when it lives Hunter's canal and the first portion of popliteal artery. Intermuscular vastoadductoria sept is dissected and the following arteries are ligated and dissected: а. superior medialis genus, а. superior lateralis genus.
  Interventions: Procedure: Angioplasty with stenting of the femoral artery, supplemented by fasciotomy in Hunter's channel

INTERVENTIONS:
Procedure: Angioplasty with stenting of the femoral artery — A standard endovascular exposure is carried out under local anesthesia and a lesioned arterial segment is visualized. Stenosis or artery occlusion is passed by the hydrophilic guide. During the occlusion transluminal or subintimal artery recanalization (most frequently mixed) is conduced. Then balloon angioplasty of stenosis or occlusion are carried out. After the angiographic control if necessary stent (balloon extpandable or self-expanding) of all the extension is mounted.
  Medical therapy includes aspirin (acid acetylsalicylic) prescription before the procedure (160 - 300 mg/d), beginning from minimum per day and heparin (heparin sodium) injection during the procedure (5000 U iv). After the procedure aspirin (acid acetylsalicylic) in dose 100 mg/d within long period should be prescribed in all the patients, and plavix (clopidogrel) in dose 75/d should be prescribed within 3 months.
  Arms: Stenting of the femoral artery.
Procedure: Angioplasty with stenting of the femoral artery, supplemented by fasciotomy in Hunter's channel — Standard endovascular stenting of femoral artery. The exposure is carried out to the distal part of superficial femoral artery when it lives Hunter's canal and the first portion of popliteal artery. Intermuscular vastoadductoria sept is dissected and the following arteries are ligated and dissected: а. superior medialis genus, а. superior lateralis genus.
  Medical therapy includes aspirin (acid acetylsalicylic) prescription before the procedure (160 - 300 mg/d), beginning from minimum per day and heparin (heparin sodium) injection during the procedure (5000 U iv). After the procedure aspirin (acid acetylsalicylic) in dose 100 mg/d within long period should be prescribed in all the patients, and plavix (clopidogrel) in dose 75/d should be prescribed within 3 months.
  Arms: Stenting of the femoral artery and fasciotomy.

SUMMARY:
Comparison of two methods for revascularization of the superficial femoral artery: stenting of the superficial femoral artery vs. stenting of the superficial femoral artery supplemented with fasciotomy in Hunter canal in patients with steno-occlusive lesion of the femoro-popliteal segment of TASC C, D.

DETAILED DESCRIPTION:
Physiological flexions and extensions in hip and knee joints cause dramatic deformity in stented femoral and superficial femoral arteries, both axially and angularly. As a result, stents get broken, restenosed or thrombosed. Some researchers report a 20 to 46% two-year incidence of broke stents in the superficial femoral artery, while restenosis and occlusion incidence vary from 21.8% to 53.3% . In addition to axial and angular stress, contributing to this untoward effect is musculofascial sheath which houses the artery in distal thigh.

Investigators suggest that standard stenting of an artery be augmented by incision of the anterior musculofascial sheath (septum intermuscular vastoadductoria) that will increase the mobility of distal part of the femoral artery, which will decrease frequency breakage of stents. Review of the world literature yielded no peer instances of such improvement of stenting outcomes in the said arteries.

ELIGIBILITY:
Inclusion Criteria:

* Patients with occlusive lesions of C and D type iliac segment, and with chronic lower limb ischemia (II-IV degree by Fontaine, 4-6 degree by Rutherford).
* Patients who consented to participate in this study.

Exclusion Criteria:

* Chronic heart failure of III-IV functional class by NYHA classification.
* Decompensated chronic "pulmonary" heart
* Severe hepatic or renal failure (bilirubin> 35 mmol / l, glomerular filtration rate <60 mL / min);
* Polyvalent drug allergy
* Cancer in the terminal stage with a life expectancy less than 6 months;
* Acute ischemic
* Expressed aortic calcification tolerant to angioplasty
* Patients with significant common femoral artery lesion
* Patient refusal to participate or continue to participate in the study

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-10 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Ankle-brachial index | Baseline, 3 days after the operation, 6 month, 12 month, 2 years
  Change in ankle-brachial index.
Ultrasound scan of the operated segment | Baseline, 3 days after the operation, 6 month, 12 month, 2 years
  The degree of stenosis in the operated segment.
CT-angiography of lower limb arteries | Baseline, 3 days after the operation, 6 month, 12 month, 2 years
  The degree of stenosis in the operated segment. CT-angiography of lower limb arteries at the control points will be done only if the detection of steno-occlusive lesions of the operated segment during the observation period, confirmed by ultrasound.

SECONDARY OUTCOMES:
Number of participants with a successful procedure of revascularization. | During the operation.
  Number of participants with a successful procedure of revascularization.
Number of participants with complications during the operation. | During the operation.
  Number of participants with complications during the operation.
Number of participants with limb salvage | 3 days after the operation, 6 month, 12 month, 2 years
  Number of participants with limb salvage.

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Karpenko, Study Director — Scientific-Research Institute of Circulation Pathology named after Academician E. Meshalkin
Locations (1):
- NRICP, Novosibirsk, Russia

REFERENCES:
- [Derived] Karpenko AA, Rabtsun AA, Popova IV, Saaya SB, Gostev AA, Ignatenko PV, Starodubtsev VB, Cheban AV. Influence of lamina vastoadductoria dissection on the outcomes of femoral artery extensive lesion stenting: A pilot randomised investigation. J Biomech. 2022 May;136:111053. doi: 10.1016/j.jbiomech.2022.111053. Epub 2022 Mar 19. PMID 35366499